CLINICAL TRIAL: NCT01831232
Title: Idarubicin, Cytarabine and Pravastatin (IAP) for Induction of Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: Idarubicin, Cytarabine, and Pravastatin Sodium in Treating Patients With Acute Myeloid Leukemia or Myelodysplastic Syndromes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mazyar Shadman, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2674.00; NCI-2013-00743 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2674.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2013-04-08; First posted 2013-04-15 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Refractory Anemia With Excess Blasts; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Anemia, Refractory, with Excess of Blasts | interventions — Pravastatin; Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (pravastatin sodium, idarubicin, and cytarabine) (Experimental): Patients receive pravastatin sodium PO QD on days 1-8, idarubicin IV over 10-15 minutes on days 4-6, and cytarabine IV continuously on days 4-7. Treatment repeats every 28-56 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pravastatin sodium; Drug: idarubicin; Drug: cytarabine; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: pravastatin sodium — Given PO
  Other Names: PRAV; Pravachol
Drug: idarubicin — Given IV
  Other Names: 4-demethoxydaunorubicin; 4-DMDR; DMDR; IDA
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies idarubicin, cytarabine, and pravastatin sodium in treating patients with newly diagnosed acute myeloid leukemia or myelodysplastic syndromes. Drugs used in chemotherapy, such as idarubicin and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Pravastatin sodium may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving idarubicin and cytarabine together with pravastatin sodium may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the rate of achieving a "good complete response (CR)" after treating patients with newly diagnosed acute myeloid leukemia (AML) with idarubicin, cytarabine and pravastatin (pravastatin sodium) (IAP).

II. To determine the toxicity (death within 28 days of starting therapy = treatment related mortality or "TRM") with IAP in newly-diagnosed AML.

SECONDARY OBJECTIVES:

I. To determine rates of complete remission (CR), remission with incomplete blood count recovery (CRi), partial remission (PR), relapse-free survival and overall survival.

II. To identify biomarkers (ie. changes in serum cholesterol) associated with clinical responses.

OUTLINE:

Patients receive pravastatin sodium orally (PO) once daily (QD) on days 1-8, idarubicin intravenously (IV) over 10-15 minutes on days 4-6, and cytarabine IV continuously on days 4-7. Treatment repeats every 28-56 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then annually for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of acute myeloid leukemia by World Health Organization (WHO) 2008 criteria, including patients with >= 20% blasts in the bone marrow or peripheral blood (except acute promyelocytic leukemia), or myelodysplastic syndrome refractory anemia with excess blasts (RAEB)-2 by WHO classification or advanced myeloproliferative neoplasm with >= 10% blasts in the bone marrow or peripheral blood, including chronic myelomonocytic leukemia (CMML) CMML-2 by WHO 2008 classification
* Untreated AML or high-risk myelodysplastic syndrome (MDS) and a simplified TRM score of =< 9.2
* Bilirubin < 2.0 mg/ml
* Any creatinine value is acceptable
* Any performance status is eligible
* Life expectancy otherwise > 1 year
* Patients are not excluded based on cardiac history
* Females of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment
* Patients must use an effective contraceptive method during the study and for a minimum of 90 days after study treatment
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mazyar Shadman, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pravastatin Sodium, Idarubicin, and Cytarabine)
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pravastatin Sodium, Idarubicin, and Cytarabine)
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 57 [35 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 9
Diagnosis [Count of Participants; unit: Participants]
  Acute Myeloid Leukemia (AML) | 21
  Myelodysplastic Syndrome (MDS) | 2
  Chronic Myelomonocytic Leukemia (CMML) | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Good Complete Remission (CR)
Description: A Bayesian design intended to simultaneously monitor efficacy and toxicity will be used.
  Definition of Good CR: Conventional criteria for CR (absolute neutrophil count > 1,000/uL, platelet count > 100,000/uL, marrow with <5% morphologic blasts) and additionally the requirements that marrow Minimal Residual Disease (MRD) - detected by 10-color flow cytometry or conventional cytogenetic evaluation - be absent and that the above blood counts be obtained.
Time Frame: 35 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pravastatin Sodium, Idarubicin, and Cytarabine)
Number analyzed (Participants) | 24
Participants | 12

2. Primary Outcome: Number of Participants With TRM.
Description: A Bayesian design intended to simultaneously monitor efficacy and toxicity will be used.
  TRM: Treatment Related Mortality
Time Frame: 28 days
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Treatment (Pravastatin Sodium, Idarubicin, and Cytarabine)
Number analyzed (Participants) | 24
participants | 2 [1 to 27]

3. Secondary Outcome: Progression Free Survival (PFS)
Time Frame: 1 year after treatment with IAP
Population: Patients who had a good complete remission (CR), CR with evidence of minimal residual disease (MRD), or complete remission with incomplete blood count recovery (CRi) following treatment. Cheson AML Response Criteria are used to assess response.Good CR is defined as <5% blasts in marrow, no MRD and recovery of blood counts by day 35 after induction.
Measure: Number (95% Confidence Interval); unit: percentage of patients with PFS
Arm/Group | Treatment (Pravastatin Sodium, Idarubicin, and Cytarabine)
Number analyzed (Participants) | 17
percentage of patients with PFS | 52.6 [28.7 to 71.9]

4. Secondary Outcome: Overall Survival
Description: Amount of time a patient lives after treatment with IAP
Time Frame: 1 year after treatment with IAP
Measure: Number (95% Confidence Interval); unit: percentage of patients surviving
Arm/Group | Treatment (Pravastatin Sodium, Idarubicin, and Cytarabine)
Number analyzed (Participants) | 24
percentage of patients surviving | 53.5 [32 to 71]

5. Secondary Outcome: Number of Biomarker-positive Participants With Clinical Responses
Description: Biomarkers: FLT3-ITD positive, NPM1 positive, CEBPA. A "good CR" is defined as <5% blasts in the marrow by morphologic evaluation along with the absence of any MRD by flow cytometry or cytogenetics and recovery of blood counts (platelets >100,00 and absolute neutrophil count >1,000) by day 35 after induction. Cheson AML Response Criteria is used for Morphologic Leukemia Free State, Morphologic Complete Remission, Cytogenetic Complete Remission (CRc), Molecular Complete Remission (CRm), Morphologic Complete Remission with Incomplete Blood Count Recovery (CRi), Partial Remission (PR), Treatment Failure, Recurrence (Progressive Disease).
Time Frame: 38 days after dosing
Population: Participants with biomarkers: FLT3-ITD positive, NPM1 positive or CEBPA
Measure: Number; unit: participants with clinical responses
Arm/Group | Treatment (Pravastatin Sodium, Idarubicin, and Cytarabine)
Number analyzed (Participants) | 6
participants with clinical responses | 0

6. Secondary Outcome: Rate of Complete Remission (CR), Remission With Incomplete Blood Count Recovery (CRi) and Partial Remission (PR)
Description: Complete remission (CR) - includes patients with good CR and CR with minimal residual disease (MRD); remission with incomplete blood count recovery (CRi), partial remission (PR)
Time Frame: 35 days
Population: All patient who received IAP treatment were assessed for response. The number of participants with CR, CRi and PR are included in the table below.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pravastatin Sodium, Idarubicin, and Cytarabine)
Number analyzed (Participants) | 24
Participants
  CR | 15
  CRi | 2
  PR | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Pravastatin Sodium, Idarubicin, and Cytarabine)
All-Cause Mortality (participants affected / at risk) | 6/24
Serious Adverse Events (participants affected / at risk) | 2/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pravastatin Sodium, Idarubicin, and Cytarabine) (N=24)
Multi organ failure secondary to sepsis (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pravastatin Sodium, Idarubicin, and Cytarabine) (N=24)
Febrile neutropenia Grade 3 (Blood and lymphatic system disorders) | 17 (17)
Febrile neutropenia Grade 4 (Blood and lymphatic system disorders) | 1 (1)
Rash Grade 3 (Skin and subcutaneous tissue disorders) | 3 (3)
Hand-foot syndrome Grade 3 (Skin and subcutaneous tissue disorders) | 2 (2)
Septic shock (Grade 4) (Infections and infestations) | 1 (1)
Diarrhea Grade 3 (Gastrointestinal disorders) | 6 (6)
Nausea/Vomiting (Gastrointestinal disorders) | 4 (4)
Mucositis (Gastrointestinal disorders) | 3 (3)
Transaminitis Grade 3 (Investigations) | 2 (2)
Colon pneumatosis Grade 3 (Gastrointestinal disorders) | 1 (1)
GI bleeding Grade 3 (Gastrointestinal disorders) | 1 (1)
Tumor lysis syndrome Grade 3 (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No